CLINICAL TRIAL: NCT03874286
Title: The Together Project-Transplant Organ Genomics to Help Prevent Rejection in Liver Transplant Recipients
Brief Title: The TOGETHER Project - Liver
Acronym: TOGETHER
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark Stegall, Principal Investigator, Mayo Clinic
Other Study IDs: IRB# 16-006453
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Liver Transplant Rejection
Keywords: Liver Transplant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Any unused specimens will be destroyed or stored at Mayo Clinic. Peripheral blood obtained under this protocol may be used in future assays to reevaluate biological responses as additional research tests are developed or refined over time. Samples may be used to look at genetic information in relation to liver transplantation (for example, the rejection process). However, samples could also be used in studies that are not related to transplantation (for example, the immune system as a whole).
  Specimens will not be stored for longer than 15 years after the closure of the study. Appropriate informed consent will be obtained for both the collection and storage of samples. Any future research identified will be reviewed and approved by an Institutional Review Board.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver Transplant: Participants will obtain a liver biopsy at 4 months post transplant and 12 months post transplant.
  Interventions: Diagnostic Test: Liver Transplant

INTERVENTIONS:
Diagnostic Test: Liver Transplant — Patients will obtain a research blood draw and a liver biopsy at 4 months and 12 months post transplant. Liver biopsies are routinely performed in the liver transplant population. We will be obtaining a liver biopsy at this particular time point to compare the biopsy results with the peripheral blood results.
  Other Names: Liver biopsy

SUMMARY:
To validate the use of a RNAseq-based peripheral blood assay in liver transplant recipients when correlated to liver biopsy results.

DETAILED DESCRIPTION:
The study is a prospective, observational study utilizing peripheral blood assays that will be collected at time points that are considered standard of care at most institutions. 100 participants will be enrolled in study. Participants will have peripheral blood collected at 4 months and 12 months after liver transplant, as well as any for cause time points. Participants will also have liver biopsies collected at these time points. The results from the liver biopsies will be used in correlation with the results from the peripheral blood assays.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given informed consent and are willing to comply with the protocol, including the use of their peripheral blood specimens and data for subsequent research.
* Patients with increased risk of rejection. Patients must meet at least one of the following criteria:

  1. Autoimmune etiology of the original liver disease (autoimmune hepatitis, primary biliary cirrhosis or primary sclerosing cholangitis)
  2. Recipients of donation-after-cardiac death (DCD) donors
  3. Recipients of simultaneous liver-kidney transplantation
  4. Positive crossmatch liver transplant (T cell flow crossmatch or B cell flow crossmatch).

     Exclusion Criteria:
* Adult ( ≥ = 18 years) renal transplant recipient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult liver transplant recipients with diverse demographics (e.g. recipient race and donor type) and treatment strategies (induction, steroid-free, etc.).
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
To validate the use of a RNAseq-based peripheral blood assay in liver transplant recipients when correlated to liver biopsy results. | 3 years
  The primary endpoint for this study is defined as obtaining the results of the RNAseq testing and to determine if an assay for rejection can be developed.

SECONDARY OUTCOMES:
To validate the use of a RNAseq-based peripheral blood assay in liver transplant recipients when correlated to liver biopsy results. | 3 years
  The secondary endpoint for this study is defined as obtaining the results of the RNAseq testing and to ascertain whether an assay for detection of disease recurrence can be developed.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stegall, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials